CLINICAL TRIAL: NCT03507218
Title: Clinical, Laboratory, and Biomedical Characterization of Pediatric Acute-onset Neuropsychiatric Syndrome (PANS)
Brief Title: Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS)
Status: Terminated | Type: Observational
Why Stopped: PI left and section closed.
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180036; 18-M-0036
Record Dates: First submitted 2018-04-24; First posted 2018-04-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Pediatric Acute-onset Neuropsychiatric Syndrome (PANS)
Keywords: Obsessive Compulsive Disorder; Anxiety Disorder; PANDAS (Pediatric Autoimmune Neuropsychiatric Disorders Associated d; Eating Disorders
MeSH Terms: conditions — Pediatric acute-onset neuropsychiatric syndrome; Obsessive-Compulsive Disorder; Anxiety Disorders; Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Children with Pediatric Acute-onset Neuropsychiatric Syndrome (PANS)

SUMMARY:
Background:

PANS is an illness that comes on suddenly in children. The full name is Pediatric Acute-Onset Neuropsychiatric Syndrome. It can cause sudden obsessive-compulsive behaviors. It can also cause children to suddenly restricte their food intake. Researchers want to learn more about children with PANS. They also want to learn more about the illness.

Objective:

To study some disorders of behavior and emotion that start in childhood.

Eligibility:

Children 3 14 years old who have had severe obsessive-compulsive symptoms or food restriction start quickly

Design:

Parents will answer questions. The topics include:

Their child s medical history

Their child s physical and mental health

Their family history. The focus will be on neurodevelopmental and psychiatric conditions. A family tree will be drawn.

Participants will have a physical exam.

Participants may take tests on paper or computer. These will focus on thinking, memory, and behavior.

Participants and parents will give a blood sample.

Participants will have magnetic resonance imaging (MRI). A strong magnetic field and radio waves take pictures of the brain. Participants will lie on a table that slides in and out of a metal scanner.

Participants may have photos or videos taken.

Participants may have other tests. These may include heart tests, sleep tests, and lumbar puncture.

Sponsoring Institute: National Institute of Mental Health

DETAILED DESCRIPTION:
This multi-site study is intended to collect data and samples from a nationwide cohort of children with Pediatric Acute-onset Neuropsychiatric Syndrome (PANS). PANS is defined by three clinical criteria:

1. Abrupt, dramatic onset of obsessive-compulsive disorder (OCD) or severely restricted

   food intake AND
2. Concurrent presence of additional neuropsychiatric symptoms, with similarly severe and acute onset, from at least two of the following seven categories:

   * Anxiety (particularly separation anxiety)
   * Emotional lability and depression
   * Irritability, aggression, and/or severely oppositional behaviors
   * Behavioral (developmental) regression
   * Deterioration in school performance (due to inattention, concentration difficulties, memory deficits, or others)
   * Sensory or motor abnormalities
   * Somatic signs and symptoms, including sleep disturbances, enuresis, or urinary frequency
3. Symptoms are not better explained by a known neurologic or medical disorder, such as Sydenham chorea, systemic lupus erythematosus, Tourette disorder, or others.

As a clinical syndrome, PANS likely represents a number of different disorders with unique symptom constellations, disease mechanisms, and etiologies. The purpose of this investigation is to identify these distinctive disorders by carefully documenting, archiving, and analyzing the clinical features of each case of PANS, including not only details of the onset and course of symptoms, but also results of physical examination, laboratory assays, and paraclinical assessments, such as electroencephalography (EEG), polysomnography (PSG), brain imaging (e.g., magnetic resonance imaging [MRI] scans), and others. In addition to defining the unique clinical features associated with a specific disorder, we also hope to identify biomarkers of risk and disease severity, including not only determinant genes, but also environmental triggers, such as those producing post-infectious autoimmunity (e.g., Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infection, or PANDAS). To accomplish this, we propose to collect and archive clinical information and biospecimens at different stages of the illness (e.g., initial onset, first exacerbation, following known environmental triggers, during convalescence, etc.) and also to compare these results against data and specimens obtained from healthy controls and children with non-PANDAS OCD, tics, anxiety disorders, or eating disorder. Clinical, laboratory, and biomedical data will be stored in the NIMH database (housed on the Clinical Trials Database [CTDB] of NICHD) and blood, genetic material, and other biospecimens, including microbial cultures, stored in the NIMH Genetics/Biological Repository. There are two types of baseline evaluations within this protocol. The first is limited to participants with acute-onset neuropsychiatric symptoms (PANS subjects) and will be conducted in the NIH Clinical Center by investigators from the NIMH Section on Behavioral Pediatrics (Drs. Swedo, Grant, and Hommer.) These in-depth phenotyping evaluations will include medical and psychiatric history, family history, completion of standardized questionnaires, physical and neurological examinations, neuropsychological testing, MRI scan, throat swab (for microbiologic testing), cheek swab (to obtain genetic samples), and phlebotomy to obtain blood for laboratory assays and genetic testing. Children with undiagnosed acute-onset neuropsychiatric symptoms may undergo additional testing as part of the diagnostic evaluation; these assessments might include (among others), electroencephalography (EEG), echocardiogram/electrocardiogram (ECHO/ECG) and/or polysomnography (PSG). If the child s clinical presentation warrants a lumbar puncture as part of the diagnostic evaluation, (e.g. abnormal findings on neurologic exam, EEG or PSG, or lab abnormalities suggestive of systemic autoimmunity or neuroinflammation), a sample of cerebrospinal fluid will be collected for research, as well as for clinical testing. Sedation will not be used for these lumbar punctures, nor will it be used for any research purposes in this protocol.

The second type of baseline evaluation will be used at NIMH for subjects with non-PANDAS psychiatric disorders and healthy volunteers. At participating extramural institutions, this is the evaluation that will be used for all participants (PANS, non-PANS, healthy volunteers) evaluated. These evaluations will include standardized questionnaires, medical and psychiatric history, family history, physical examination, throat swab (for microbiologic testing), cheek swab (to obtain genetic samples), and phlebotomy to obtain blood for clinical assays and research, including genetic studies. The assessments will generally be completed in an outpatient clinic at the participating site, but also might be performed on hospitalized children, if their medical condition permits research participation. Family members of PANS probands will have a medical and psychiatric history and physical exam and provide a blood sample (or cheek swab) for genetic research.

The Affected Probands, Healthy Volunteers, and Subjects with Non-PANS Psychiatric Disorders will have follow-up evaluations annually, as well as on Ad Hoc basis. The Annual check-ups will include an interim clinical history and relevant symptom ratings (tailored to the subject s clinical profile). These follow-up evaluations may be done by phone or videoconference. Ad hoc evaluations will occur during periods of health (if not healthy at baseline) and during an episode of acute illness (either infectious illness or neuropsychiatric symptom exacerbations) and convalescence (at least 8 weeks after recovery). These in-person evaluations will include an interim clinical history, relevant symptom ratings, phlebotomy to obtain research bloods, and in some cases, acquisition of microbial samples (oral, nasal, nasopharyngeal and/or pharyngeal swabs, and feces). To identify biomarkers of disease and recovery, children with PANS may be followed until their 18th birthday, even if fully recovered from their acute illness. Healthy volunteers and psychiatric controls will be followed no longer than 3 years from study entry.

This is a natural history study, with the primary goal of collecting clinical data and biospecimens in order to identify subgroups of patients sharing a common disease mechanism and thus provide opportunities for development of new treatment and prevention strategies. The wealth of clinical information and the large number of biologic and genetic samples acquired in this prospective, longitudinal investigation also permits us to address four specific aims:

1. Identify unique and distinctive clinical, paraclinical, and laboratory features of acuteonset neuropsychiatric disorders among patients meeting criteria for PANS.
2. Determine the role of environmental pathogens, such as Group A streptococci, in the etiopathogenesis of acute-onset neuropsychiatric disorders.
3. Investigate factors influencing host susceptibility and resistance.
4. Elucidate the role of immune dysfunction in PANS or a subgroup of its patients.
5. Provide clinical diagnostic assessments to children with undiagnosed acute-onset neuropsychiatric symptoms.

ELIGIBILITY:
* INCLUSION CRITERIA:

Affected Probands (Children with PANS) will be eligible if they:

1. Are 3 to 14 years of age (initial enrollment must occur prior
2. Have a history of abrupt onset (less than 24-48 hours) of impairing OCD and/or eating restrictions.
3. Are able to travel safely to the regional medical center where the evaluations will be conducted and are able to be examined safely over a period of one or more days.
4. Assent to participate (if they are at least seven years old and have capacity to do so) and have legal guardians who consent to their minor child s participation.
5. Are under the care of a primary physician in their home community.

First-degree Relatives will be eligible if they:

1. Are a biologic parent or sibling of an affected proband.
2. Consent (or assent) to undergo study evaluations and to provide blood, microbial and genetic samples.

Children with Non-PANS Neuropsychiatric Symptoms may be enrolled if they:

1. Are 3 to 14 years of age (initial enrollment must occur prior to the participant s 15th birthday to permit prospective longitudinal evaluations)
2. Have OCD, tics, anxiety disorders, or other psychiatric symptoms, but do NOT have a history of acute symptom onset.
3. Are willing to participate in medical, psychiatric, and behavioral assessments and to provide bio-specimens including blood, urine, and microbial flora (mouth, oropharynx, and/or stool).
4. Assent to participate (if they are at least seven years old and have capacity to do so) and have legal guardians who consent to their minor child s participation.
5. Are under the care of a primary physician in their home community.

Healthy Pediatric Volunteers may be enrolled if they:

1. Are 3 to 14 years of age (initial enrollment must occur prior to the participant s 15th birthday to permit prospective longitudinal evaluations).
2. Are physically healthy and do not have psychiatric symptoms.
3. Are willing to participate in medical, psychiatric, and behavioral assessments and to provide bio-specimens including blood, urine, and microbial flora (mouth, oropharynx, and/or stool).
4. Assent to participate (if they are at least seven years old and have capacity to do so) and have legal guardians who consent to their minor child s participation.

EXCLUSION CRITERIA:

Participants will not be eligible if they:

1. Appear to the investigators to be too unstable psychiatrically or medically to participate safely in the protocol.
2. Are unwilling or unable to be evaluated and followed prospectively.
3. Have a parent/guardian who is not willing to participate at a distance through web-based or phone-based data collection.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: study population will include potential participants from primary care and specialty medical referrals, community samples, and self-referral from across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Establish national database and samples repository for pediatric acute-onset neuropsychiatric syndrome (PANS) | Study Completion

SECONDARY OUTCOMES:
Identify unique and distinctive features of subgroups of patients with PANS, in order to determine the shared disease mechanism | Study completion
Elucidate the role of immune dysfunction in the syndrome of PANS, as well as for subgroups of patients | Study completion
Determine role of environmental pathogens, such as Group A streptococci, in the etiopathogenesis of PANS | Study completion
Investigate factors influencing host susceptibility and resistance | Study completion

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Swedo, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (8):
- United States (8):
  - University of Arizona, Tucson, Arizona
  - Lucille Salter Packer Children's Hospital, Stanford, California
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - University of Southern Florida, Tampa, Florida
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Harvard Medical School, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri

REFERENCES:
- [Background] Chang K, Frankovich J, Cooperstock M, Cunningham MW, Latimer ME, Murphy TK, Pasternack M, Thienemann M, Williams K, Walter J, Swedo SE; PANS Collaborative Consortium. Clinical evaluation of youth with pediatric acute-onset neuropsychiatric syndrome (PANS): recommendations from the 2013 PANS Consensus Conference. J Child Adolesc Psychopharmacol. 2015 Feb;25(1):3-13. doi: 10.1089/cap.2014.0084. Epub 2014 Oct 17. PMID 25325534
- [Background] Williams KA, Swedo SE. Post-infectious autoimmune disorders: Sydenham's chorea, PANDAS and beyond. Brain Res. 2015 Aug 18;1617:144-54. doi: 10.1016/j.brainres.2014.09.071. Epub 2014 Oct 7. PMID 25301689